CLINICAL TRIAL: NCT02773836
Title: European Regulatory Science on Tobacco: Policy Implementation to Reduce Lung Diseases (EUREST-PLUS)
Acronym: EUREST-PLUS
Status: Completed | Type: Observational
Sponsor: European Network For Smoking and Tobacco Prevention (Other)
Collaborators: King's College London (Other); German Cancer Research Center (Other); Maastricht University (Other); University of Athens (Other); AER PUR ROMANIA (Unknown); European Respiratory Society (Other); University of Waterloo (Other); Institut Català d'Oncologia (Other); DOHANYZAS VAGY EGESZSEG MAGYAR ALAPITVANY (Unknown); PROMOCJA ZDROWIA - ZDROWIE ALBO TYTON FUNDACJA (Unknown); University of Crete (Other); TNS OPINION SA (Unknown)
Responsible Party: Sponsor
Other Study IDs: 681109
Record Dates: First submitted 2016-05-11; First posted 2016-05-16 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Tobacco Dependence
Keywords: tobacco use; e-cigarettes; public policy; ITC
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use; Vaping | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Greek cohort: Participants recruited from Greece will receive a questionnaire at pre- and post- intervention
  Interventions: Other: Questionnaire
- German cohort: Participants recruited from Germany will receive a questionnaire at pre- and post- intervention
  Interventions: Other: Questionnaire
- Romanian Cohort: Participants recruited from Romania will receive a questionnaire at pre- and post- intervention
  Interventions: Other: Questionnaire
- Spanish Cohort: Participants recruited from Spain will receive a questionnaire at pre- and post- intervention
  Interventions: Other: Questionnaire
- Hungarian Cohort: Participants recruited from Hungary will receive a questionnaire at pre- and post- intervention
  Interventions: Other: Questionnaire
- Polish cohort: Participants recruited from Poland will receive a questionnaire at pre- and post- intervention
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)

SUMMARY:
The main objective of EUREST-PLUS is to monitor and evaluate the impact of the Tobacco Products Directive (TPD) within the context of FCTC ratification at an EU level. The investigators specific objectives, within WorkPackage 2 and Workpackage 3 are: To evaluate the psychosocial and behavioral impact of TPD implementation and FCTC implementation, through the creation of a cohort study of adult smokers in 6 European Member States (EU MS), Germany, Greece, Hungary, Poland, Romania, Spain; (total n=6000) in a pre- vs. post-TPD study design.

EUREST-PLUS is funded through the European Union's Horizon 2020 research and innovation programme under grant agreement No 681109

DETAILED DESCRIPTION:
Smoking and other forms of tobacco consumption are considered the single most important cause of preventable morbidity and premature mortality worldwide, with tobacco the major single cause for premature deaths in the European Union (EU).Efforts to reduce the devastation of tobacco-related deaths and illness in the EU consist of its newly adopted binding legislation, the Tobacco Products Directive (TPD), and the ongoing implementation of the WHO Framework Convention on Tobacco Control (FCTC).

Objective:

The main objective of EUREST-PLUS is to monitor and evaluate the psychosocial and behavioral impact of the TPD within the context of FCTC ratification at a European level, through the creation of a cohort study of adult smokers in 6 EU MS (Germany, Greece, Hungary, Poland, Romania, Spain; total n=6000) in a pre- vs. post-TPD study design. The baseline recruitment will take place in WP2 and the follow up in WP3.

Sampling frames:

* The sampling frame will be determined through a national probability sampling design within each country.
* Sample stratification will be geographic and comprise the major regions of each country (Nomenclature of Territorial Units for Statistics - NUTS) NUTS2 (Basic regions for the application of regional policies) will be used for all countries except Germany - where NUTS1 (Major socio-economic regions) will be used, as well as degrees of urbanization (city/town/rural.)
* Geographic areas excluded from the sampling design will be: In Greece, the islands in the Ionian Sea, the northern Aegean Sea and the southern Aegean Sea. In Spain the Canaries, Ceuta and Melilla
* Overall the design will be multistage within strata. The strata will be conceptually divided into clusters, each the size of an enumeration area, with the objective of sampling a total of 250 clusters - 4 adult smokers per cluster in every country.
* Clusters will be allocated based on population size and sampled via random sampling.

Sampling households within clusters:

* Interviewers will employ a random walk procedure within a particular cluster
* Once interviewers have arrived at an address, the household will be approached four times at different times of the day and week before being designated as "unable to be contacted."
* If an address corresponds to multiple households, a single household will be chosen at random.
* Households are approached until a total of 4 adult smokers have been reached within the cluster. A maximum of one male smoker and one female smoker will be selected for interview in each household.
* One male and one female from within the household that meet the criteria will be selected using the last birthday method

Respondents:

* The respondents for the Survey will be smokers aged 18 and older. The first part of the survey, which is the household screener, contains the questions that are used to determine whether the household has members that meet the criteria for inclusion.

  * The household screener is asked of the most knowledgeable individual (MKI) within the household.
  * One male and one female from within the household that meet the criteria will be selected using the last birthday method.
* The Individual screener follows the Household screener and confirms the information from the MKI is accurate. If the selected individual meets the eligibility criteria and consents to participate, they will be included in the sample

Survey (questionnaire):

The questionnaire will include questions not only about tobacco use, history of use, history of quitting, quit method(s) used, measures of dependence, and demographics (age, gender, education, income) but also extensive, theory-based measures of responsiveness to each policy domain of the FCTC. The survey questionnaire will consist of:

1. multiple measures of policy-specific variables for each of the domains of the TPD and FCTC (e.g., health warnings, additives, e-cigarettes for TPD, illicit trade; additional domains of the FCTC, including smoke-free laws, tax/price policies, cessation services, additional product regulation domains);
2. psychosocial mediators, identified by past research and theory to predict future health behaviours, including beliefs and attitudes, perceived risk, intentions to quit;
3. moderators such as demographic variables (sex, gender), and other variables that will allow analyses of whether TPD and FCTC policies vary in their impact as a function of socioeconomical status.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Must smoke at least monthly.
* Must have smoked 100 cigarettes in their lifetime.
* Must live in the household visited

Exclusion Criteria:

* Inability to complete the questionnaire due to health/mental incapability.
* Unable to provide consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of 1,000 smokers recruited in each of 6 European Member States (n=6,000 in total), to be recruited at baseline.
Sampling Method: Probability Sample
Enrollment: 6036 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2018-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Vardavas, MD,RN,MPH,PHD, Principal Investigator — European Network For Smoking and Tobacco Prevention
Locations (1):
- European Network For Smoking and Tobacco Prevention, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The reason there are more participants enrolled at Period 2 (Wave 2 Post-TPD implementation) as compared to Period 1 (Wave 1 Pre-TPD implementation) is because a replenishment sample was recruited in Wave 2.
Groups:
- Greek Cohort: Participants recruited from Greece
  Questionnaire: Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)
- German Cohort: Participants recruited from Germany
  Questionnaire: Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)
- Romanian Cohort: Participants recruited from Romania
  Questionnaire: Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)
- Spanish Cohort: Participants recruited from Spain
  Questionnaire: Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)
- Hungarian Cohort: Participants recruited from Hungary
  Questionnaire: Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)
- Polish Cohort: Participants recruited from Poland
  Questionnaire: Questionnaire: To evaluate the impact of the implementation of the EU Tobacco Products Directive (TPD) and Framework Convention on Tobacco Control (FCTC)
Period: Wave 1- Pre-TPD Implementation
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Started | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Completed | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wave 2- Post-TPD Implementation
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Started (The reason there are more participants in Period 2 is because a replenishment sample was also used) | 1010 | 1013 | 1003 | 1010 | 1002 | 998
Completed | 1010 | 1013 | 1003 | 1010 | 1002 | 998
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort | Total
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006 | 6011
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 888 | 903 | 921 | 932 | 898 | 900 | 5442
  >=65 years | 112 | 100 | 80 | 69 | 102 | 106 | 569
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.5) | 45.5 (14.6) | 43.9 (14.2) | 43.3 (14.4) | 46.1 (13.9) | 45.1 (14.7) | 45.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456 | 496 | 420 | 456 | 479 | 529 | 2836
  Male | 544 | 507 | 581 | 545 | 521 | 477 | 3175
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Cigarettes/E-cigarettes Smoked per day by participants [Mean (Standard Deviation); unit: cigarettes per day] — How many cigarettes/E-cigarettes do you smoke per day?
  Collected via questionnaire Cigarettes/day (all current smokers)
  cigarettes per day | 20.2 (12.8) | 14.9 (9.0) | 16.0 (8.9) | 14.9 (9.2) | 15.9 (7.4) | 15.9 (7.7) | 16.3 (9.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Think About the Harm of Smoking
Description: In the last 30 days, how often did you think about the harm your smoking might be doing to you? responses:
  1. Never
  2. Rarely
  3. Sometimes
  4. Often
  5. Very often
  8 Refused 9 Don't know
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Participants
  Never | 67 | 272 | 192 | 194 | 228 | 248
  Rarely | 139 | 265 | 103 | 172 | 295 | 260
  Sometimes | 314 | 321 | 259 | 333 | 305 | 316
  Often | 327 | 95 | 317 | 203 | 133 | 140
  Very often | 152 | 46 | 129 | 98 | 38 | 37
  Refused/ dont know | 1 | 4 | 1 | 1 | 1 | 5

2. Primary Outcome: Number of Participants Whose First Cigarette After Waking is 30 Mins or Less
Description: How soon after waking do you usually have your first smoke? responses:
  1. 5 min or less
  2. 6-30 min
  3. 31-60 min
  4. More than 60 min
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 970 | 883 | 947 | 969 | 988 | 944
Participants
  > 60 minutes | 100 | 180 | 94 | 241 | 71 | 106
  31-60 minutes | 139 | 233 | 138 | 191 | 132 | 165
  6-30 minutes | 484 | 340 | 425 | 343 | 487 | 429
  5 minutes or less | 247 | 130 | 290 | 194 | 298 | 244

3. Primary Outcome: Number of Participants Who Think About How Much They Enjoy Smoking by Frequency
Description: The following question ask you about how often you've had certain thoughts in the last 30 days. In the last 30 days, how often did you . . .
  Think about how much you enjoy smoking?
  1. Never
  2. Rarely
  3. Sometimes
  4. Often
  5. Very often
  6. Refused
  7. Don't know
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Participants
  Never | 79 | 171 | 275 | 294 | 189 | 261
  Rarely | 147 | 216 | 148 | 166 | 182 | 235
  Sometimes | 298 | 335 | 263 | 338 | 334 | 305
  Often | 325 | 197 | 220 | 150 | 247 | 143
  Very often | 149 | 65 | 92 | 53 | 44 | 50
  Refused | 0 | 0 | 0 | 0 | 0 | 4
  Don't Know | 2 | 19 | 3 | 0 | 4 | 8

4. Primary Outcome: Number of Participants Who Have Ever Tried to Quit Smoking
Description: Have you ever tried to quit smoking?
  1. Yes
  2. No
  8 Refused 9 Don't know
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Participants
  Yes | 429 | 555 | 622 | 623 | 453 | 556
  No | 571 | 448 | 379 | 378 | 547 | 447
  Refused | 0 | 0 | 0 | 0 | 0 | 3
  Don't know | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Plan to Quit Smoking
Description: Are you planning to quit smoking . . .
  1. Within the next month
  2. Within the next 6 months
  3. Sometime in the future, beyond 6 months
  4. Or are you not planning to quit?
  8 Refused 9 Don't know
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Participants
  Within the next month | 21 | 39 | 62 | 54 | 21 | 38
  Within the next 6 months | 64 | 76 | 98 | 84 | 81 | 97
  Sometime in the future, beyond 6 months | 315 | 485 | 364 | 229 | 201 | 240
  Or are you not planning to quit? | 589 | 384 | 443 | 617 | 655 | 497
  Refused | 0 | 0 | 0 | 0 | 0 | 1
  Don't know | 11 | 19 | 34 | 17 | 42 | 133

6. Primary Outcome: Number of Participants Who Think About the Harm of Smoking
Description: as for outcome 1
Time Frame: Post-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1010 | 1013 | 1003 | 1010 | 1002 | 998
Participants
  Never | 109 | 328 | 229 | 147 | 288 | 274
  Rarely | 172 | 282 | 123 | 152 | 257 | 262
  Sometimes | 393 | 248 | 264 | 407 | 310 | 299
  Often | 209 | 118 | 226 | 188 | 115 | 107
  Very Often | 127 | 36 | 158 | 116 | 30 | 53
  Don't Know | 0 | 1 | 1 | 0 | 2 | 2
  Refused | 0 | 0 | 2 | 0 | 0 | 1

7. Primary Outcome: Number of Participants Whose First Cigarette After Waking is 30 Mins or Less
Description: as for outcome 2
Time Frame: Post-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 932 | 854 | 899 | 858 | 928 | 912
Participants
  5 minutes or less | 207 | 118 | 254 | 179 | 256 | 207
  6-30 minutes | 460 | 352 | 417 | 301 | 498 | 410
  31-60 minutes | 160 | 206 | 134 | 174 | 122 | 162
  More than 60 minutes | 105 | 178 | 94 | 204 | 50 | 114
  Don't know | 0 | 0 | 0 | 0 | 2 | 19

8. Primary Outcome: Number of Participants Who Have Ever Tried to Quit Smoking
Description: Have you ever tried to quit smoking?
  1. Yes
  2. No
  8 Refused 9 Don't know
Time Frame: Post-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1009 | 1013 | 1002 | 1010 | 1000 | 991
Participants
  Has tried to quit | 367 | 505 | 553 | 517 | 431 | 475
  Never tried to quit | 581 | 444 | 364 | 370 | 518 | 468

9. Primary Outcome: Number of Participants Who Plan to Quit Smoking
Description: as for outcome 5
Time Frame: Post-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 949 | 949 | 918 | 887 | 951 | 950
Participants
  Within the next month | 11 | 26 | 46 | 39 | 19 | 12
  Within the next 6 months | 43 | 72 | 84 | 93 | 85 | 83
  Sometime in the future, beyond 6 months | 267 | 451 | 337 | 237 | 165 | 250
  Or are you not planning to quit | 613 | 390 | 422 | 509 | 648 | 497
  Refused | 3 | 0 | 0 | 0 | 0 | 0
  Don't know | 12 | 10 | 29 | 9 | 34 | 108

10. Secondary Outcome: Number of Participants Who Think About The Money They Spend on Smoking
Description: The following question ask you about how often you've had certain thoughts in the last 30 days. In the last 30 days, how often did you Think about the money you spend on smoking?
  1. Never
  2. Rarely
  3. Sometimes
  4. Often
  5. Very often
  8 Refused 9 Don't know
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Participants
  Never | 89 | 195 | 165 | 183 | 178 | 160
  Rarely | 80 | 190 | 65 | 119 | 173 | 155
  Sometimes | 205 | 284 | 166 | 297 | 284 | 346
  Often | 344 | 206 | 301 | 196 | 256 | 229
  Very often | 281 | 125 | 304 | 205 | 108 | 109
  Refused | 0 | 2 | 0 | 1 | 0 | 1
  Don't Know | 1 | 1 | 0 | 0 | 1 | 6

11. Secondary Outcome: Number of Participants Who Think About the Harm Their Smoking Might be Doing to Other People
Description: The following question ask you about how often you've had certain thoughts in the last 30 days. In the last 30 days, how often did you Think about the harm your smoking might be doing to other people?
  1. Never
  2. Rarely
  3. Sometimes
  4. Often
  5. Very often
  8 Refused 9 Don't know
Time Frame: Baseline Pre-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 1000 | 1003 | 1001 | 1001 | 1000 | 1006
Participants
  Never | 120 | 348 | 219 | 240 | 259 | 230
  Rarely | 176 | 309 | 122 | 201 | 312 | 285
  Sometimes | 302 | 259 | 261 | 319 | 274 | 315
  Often | 292 | 61 | 289 | 155 | 118 | 129
  Very often | 108 | 22 | 109 | 86 | 37 | 36
  Refused | 0 | 1 | 0 | 0 | 0 | 0
  Don't Know | 2 | 3 | 1 | 0 | 0 | 11

12. Secondary Outcome: Number of Participants Who Think About The Money They Spend on Smoking
Description: as for outcome 10
Time Frame: Post-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 949 | 949 | 918 | 887 | 951 | 950
Participants
  Never | 84 | 260 | 167 | 123 | 196 | 182
  Rarely | 98 | 184 | 57 | 115 | 210 | 161
  Sometimes | 198 | 238 | 201 | 326 | 265 | 283
  Often | 289 | 169 | 238 | 176 | 218 | 213
  Very Often | 280 | 97 | 255 | 146 | 62 | 107
  Refused | 0 | 0 | 0 | 0 | 0 | 2
  Don't know | 0 | 1 | 0 | 1 | 0 | 2

13. Secondary Outcome: Number of Participants Who Think About the Harm Their Smoking Might be Doing to Other People
Description: as for outcome 11
Time Frame: Post-TPD
Measure: Count of Participants; unit: Participants
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
Number analyzed (Participants) | 949 | 949 | 918 | 887 | 951 | 950
Participants
  Never | 114 | 367 | 225 | 157 | 307 | 277
  Rarely | 242 | 260 | 123 | 204 | 273 | 266
  Sometimes | 322 | 241 | 234 | 325 | 268 | 249
  Often | 179 | 55 | 229 | 137 | 86 | 113
  Very Often | 92 | 25 | 105 | 64 | 15 | 42
  Refused | 0 | 0 | 1 | 0 | 2 | 1
  Don't know | 0 | 1 | 1 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected
Arm/Group | Greek Cohort | German Cohort | Romanian Cohort | Spanish Cohort | Hungarian Cohort | Polish Cohort
All-Cause Mortality (participants affected / at risk) | 0/1000 | 0/1003 | 0/1001 | 0/1001 | 0/1000 | 0/1006
Serious Adverse Events (participants affected / at risk) | 0/1000 | 0/1003 | 0/1001 | 0/1001 | 0/1000 | 0/1006
Other Adverse Events (participants affected / at risk) | 0/1000 | 0/1003 | 0/1001 | 0/1001 | 0/1000 | 0/1006

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT02773836/Prot_SAP_ICF_000.pdf